**PRINCIPAL INVESTIGATOR:** Mark Roschewski, M.D.

STUDY TITLE: Phase 1 Study of Copanlisib with Dose-adjusted EPOCH-

R in Relapsed and Refractory Burkitt Lymphoma and

other High-Grade B-cell Lymphomas

STUDY SITE: NIH Clinical Center

Cohort: Screening Affected Subject

Consent Version: 02/22/2023

## WHO DO YOU CONTACT ABOUT THIS STUDY?

Principal Investigator: Mark Roschewski, M.D.

Phone: 240-760-6183

Email: mark.roschewski@nih.gov

## KEY INFORMATION ABOUT THIS RESEARCH

This consent form describes a research study and is designed to help you decide if you would like to be a part of the research study.

You are being asked to take part in a research study at the National Institutes of Health (NIH). This section provides the information we believe is most helpful and important to you in making your decision about participating in this study. Additional information that may help you decide can be found in other sections of the document. Taking part in research at the NIH is your choice.

You are being asked to take part in this study because you have relapsed and/or refractory highly-aggressive B-cell lymphomas (such as Burkitt lymphoma [BL] and certain types of diffuse large B-cell lymphoma [DLBCL]).

This consent is for "screening." We would like to find out if you are able to take part in this study.

The main purpose of this research study is to learn if it is safe to give individuals with these cancers the drug copanlisib (Aliqopa®) together with a regimen called DA-EPOCH-R which includes rituximab as well as several chemotherapy drugs. This regimen stands for dose-adjusted (**DA**), etoposide (**E**), prednisone (**P**), vincristine (**O**), cyclophosphamide (**C**), doxorubicin (**H**), and rituximab (**R**). As not every drug in this regimen is a chemotherapy, throughout this document DA-EPOCH-R will be referred to as a "combination chemotherapy regimen". We also hope to get early information if this treatment combination is an effective treatment for highly-aggressive B-cell lymphomas.

Although each is approved and used either alone or in combination to treat types of lymphoma, the use and combination of the drugs in this study is investigational. An "investigational drug" is a drug or combination of drugs that is being tested and is not approved in the United States by the U.S. Food and Drug Administration (FDA). The reason that this combination needs to be studied is to ensure that copanlisib is safe to be given with this chemotherapy regimen and that it will not be associated with any side effects that will require stopping of known effective treatment

## PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)

Version Date: 02/22/2023




such as DA-EPOCH-R. There are other drugs and treatments that may be used for your disease, and these can be prescribed by your regular cancer doctor, if you are not in this study. These drugs all work in different ways in the body as compared to the study drugs and with different side effects. If you would prefer other drugs or treatments, such as alternative chemotherapy regimens, radiation therapy, single-agent targeted therapy and/or approved forms of immunotherapy, you should consider not joining this study.

If you decide to be screened for this study, here are some of the most important things that you should know that will happen:

- We will review your health history.
- We will do physical exams, blood tests, pregnancy test, tests to look at heart function and review biopsies sample that you might have given before of your cancer and bone marrow or take new ones if tissue is not available or not done recently.
- We will review imaging tests such as a CT scan of your chest, abdomen and pelvis FDG PET/CT scan and MRI of your brain. We may need to repeat some of the scans.
- Some of the tests have risks, including risks from blood samples and contrast with the imaging. We do not know which side effects you will experience.

There may be no direct benefit to you from taking part in the study. This screening part will help us decide if you are able to take part in the next step of this research study. You will also have the benefit of seeing our NIH doctors to discuss your treatment. If you would like, we can share the results of these screening tests and notes with your personal physician.

The screening portion of this study will take between a few days and a week. If you move on to the treatment portion of the study, you may be in the study for several years depending on how you tolerate the treatment. You can stop taking part in the trial at any time.

The remaining document will now describe the research study in more detail. This information should be considered before you make your choice. Members of the study team will talk with you about the information in this document. Some people have personal, religious, or ethical beliefs that may limit the kinds of medical or research interventions in which they would want to receive participate. Take the time you need to ask any questions and discuss this study with NIH staff, and with your family, friends, and personal health care providers.

#### IT IS YOUR CHOICE TO TAKE PART IN THE STUDY

You may choose not to take part in this study for any reason. If you join this study, you may change your mind and stop participating in the study at any time and for any reason. In either case, you will not lose any benefits to which you are otherwise entitled. However, to be seen at the NIH, you must be taking part in a study or are being considered for a study. If you do choose to leave the study, please inform your study team to ensure a safe withdrawal from the research.

#### WHY IS THIS STUDY BEING DONE?

This part of the study is to determine if you are suited for the treatment part of this study.

## PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)




You may not be eligible for our study for several reasons, such as the presence of certain other diseases, infections, or problems with your organ function.

## WHAT WILL HAPPEN DURING THE STUDY?

All of these tests or procedures are part of your regular care and may be done even if you are not being considered to join the study. If you have had some of these tests or procedures recently, they may or may not have to be repeated. The tests and procedures, which may be performed as part of a separate protocol, needed to determine whether you are eligible for this trial include:

- Medical history: A complete review of your medical history, including obtaining information about your diagnosis and previous treatments, and reviewing information about your other conditions. If you have medical records from another clinic or hospital, you will be asked to get copies of these records, or your study doctor may be able to request them on your behalf.
- Physical exam: This will include taking your vital signs (temperature, blood pressure, heart rate, breathing rate), getting your height, seeing how you function in your daily activities, any current symptoms of your condition and a review of all medications that you take.
- Standard blood and urine tests:
  - o To measure your organ function, such as liver and kidney, and white blood cells, red blood cells and platelets, and blood electrolytes and blood sugars (hemoglobin A1C). Other blood tests routinely done in patients with your type of cancer will be done to confirm the status of your disease.
  - To check to see if you are pregnant if you are a woman able to get pregnant and you are not already known to be pregnant. This may be done by blood or urine test. You will not be able to participate if you are pregnant.
  - To check for cytomegalovirus (CMV) and Hepatitis B, and C infection- you will not be able to participate if you have active Hepatitis B and/or C infection or CMV as copanlisib may reactivate these viruses.
  - o To check for HIV infection: As part of this study, we will test you for infection with the human immunodeficiency virus (HIV), the virus that causes AIDS. If you are infected with HIV you may still be able to participate in this study, as long as your infection is well controlled. Your doctor may suggest medication for you to take to control your infection.

## Heart function tests:

- An electrocardiogram (EKG) will be done to check the electrical activity of your heart. An electrocardiogram (EKG) is a test that is performed while you lie still for about 5 minutes. It involves placing electrodes (small stickers that are attached to wires that go to the machine) on the chest and arms/legs and recording the electrical activity of your heart. If you have a lot of hair on your chest, it may hurt a little bit when they remove these stickers.
- An echocardiogram will test the functioning of your heart. An echocardiogram is a painless test using sound waves that takes a picture of your heart. During this test, we

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)




will put some jelly like substance on your chest. The technician will then put the ultrasound probe on your chest and record the picture. The technician may ask you to lay on your side during the test to get a better picture. For some pictures, they may put the probe on the upper part of your abdomen and push down firmly. This can be uncomfortable. The test takes about 30 minutes to complete.

- Tumor biopsy and/or tissue review: A sample of tissue from any previous surgery or biopsy of your cancer will be tested at NCI to confirm your diagnosis, stage, and status of your disease. If no tissue is available, then a biopsy will need to be performed. Usually tissue can be obtained safely and comfortably with local anesthesia. If you require conscious sedation before undergoing a biopsy, you will be informed of the risks and you will be asked to sign an additional consent prior to undergoing the procedure.
- Bone marrow testing: A bone marrow aspiration and biopsy will be done to confirm the stage and course of your disease. These are done by numbing your hipbone using a small needle containing local anesthesia, and then a needle will be put into the hipbone, and a small amount of bone marrow will be taken out through the needle.
- Imaging: Imaging to show all sites of disease, including CT scan of chest abdomen and pelvis and FDG PET/CT scan, and MRI of your brain.
  - CT (computerized tomography) scan: The CT scanner is a doughnut-shaped machine that uses x-rays to create computer pictures showing the inside of your body. During the procedure, you will need to lie still on a table inside the CT machine. The table will move you in and out of the machine during the scan and you will be instructed to hold your breath. The scan itself will only take a few minutes to complete, the entire visit will take about 30 minutes
  - o PET scans: The PET (Positron Emission Tomography) scanner is a doughnut-shaped machine that uses x-rays combined with a dose of a radioactive substance (tracer) to create computer pictures showing the inside of your body. Before the scan, you will have a radioactive substance injected into your arm after which, you will need to wait for approximately 30 minutes for the substance to be absorbed. After 30 minutes, you'll lie on a narrow, padded table and be positioned for the scan. The scan itself is painless and won't make much noise. During this time, you will need to lie very still. It will take about another 30 minutes to complete.

MRI (<u>magnetic resonance imaging</u>): MRI uses a strong magnetic field and radio waves to take pictures of the body. We will obtain pictures of your brain for this study. The MRI scanner is a metal cylinder surrounded by a strong magnetic field. During the MRI, you will lie on a table that can slide in and out of the cylinder. We will place soft padding or a coil around your head. You will be in the scanner about 45 minutes. You may be asked to lie still for up to 15 minutes at a time. While in the scanner you will hear loud knocking noises, and you will be fitted with earplugs or earmuffs to muffle the sound. You will be able to communicate with the MRI staff at all times during your scan, and you may ask to be moved out of the machine at any time.

It is very important for the experiment that you do not move your head or body inside the scanner. We will use padding around your head to help keep it in place.

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1) Version Date: 02/22/2023




We may place a bar in your mouth to help keep your head still.

#### HOW LONG WILL THE STUDY TAKE?

If you agree to take part in this study, your involvement is expected to require about a week on the screening portion. After the evaluations are complete, we will determine if you are eligible to participate in the treatment portion of the study.

## HOW MANY PEOPLE WILL PARTICIPATE IN THIS STUDY?

We plan to have approximately 39 people participate in this study at the NIH.

## WHAT ARE THE RISKS AND DISCOMFORTS OF BEING IN THE STUDY?

The primary risks or discomforts of participating in this screening are from complications caused by the tests and procedures. The following describes the most common risks of these tests and procedures. Your doctor or nurse will also discuss with you in detail any risks or discomforts of the procedures or test(s) you will be scheduled to undergo.

# Risks from tests and procedures

- Blood draws: The possible side effects of drawing blood include pain, bleeding, bruising, dizziness, light-headedness, fainting and, on rare occasions, local blood clot formation or infection with redness and irritation of the vein.
- EKG: Other than possibly experiencing some minor skin irritation from the electrodes there are no anticipated risks
- Echocardiogram: Other than the possibility of some mild discomfort during the test, there are no known risks to an echocardiogram.
- Bone marrow: The bone marrow aspiration and biopsy may cause pain, bruising, bleeding and infection. Soreness near the site may last for a couple of days after the procedure. You may have more pain, risk of bleeding and bruising if you complete both aspiration and biopsy rather than just the aspiration. If your pain is severe or you develop a fever, please contact the study team immediately.
- Tumor biopsy (if needed): The likely side effects include discomfort or pain, redness, swelling, and/or bruising at the site of the needle insertion. Bleeding from the site of the needle insertion is a less likely risk. Rarely, significant infection or bleeding from this procedure, allergic reaction to the anesthetic, or formation of a scar at the site of needle entry occurs. If you will have sedation with the procedure, these risks will be discussed with you prior to the procedure. You will be asked to sign a separate consent form prior to any biopsy procedure.
- Imaging, as applicable:
  - O CT and PET scans: There is a chance of developing an allergic reaction from the contrast material, which may cause symptoms ranging from mild itching or a rash to severe difficulty breathing, shock or rarely, death. The contrast material may also cause kidney problems. The study doctors will do a blood test prior to the test to confirm that it is safe you to receive the contrast.

## PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)




For IV contrast: You may feel discomfort when the contrast material is injected. You may feel warm, flushed, get a metallic taste in your mouth or, rarely, may make you vomit or feel sick to your stomach.

For oral contrast: You may experience vomiting, nausea, cramping, bloating, constipation or diarrhea after drinking the contrast.

See also risks from radiation below.

MRI: People are at risk for injury from the MRI magnet if they have some kinds of metal in their body. It may be unsafe for you to have an MRI scan if you have pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips (metal clips on the wall of a large artery), metal prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, tattoos, an implanted delivery pump, or shrapnel fragments. Welders and metal workers may have small metal fragments in the eye. You will be screened for these conditions before having any MRI scan. If you have a question about metal in your body, you should inform the staff. You will be asked to complete an MRI screening form before each MRI scan you have.

In addition, all magnetic objects (like watches, coins, jewelry, and credit cards) must be removed before entering the MRI scan room.

People with fear of confined spaces may become anxious during an MRI. Those with back problems may have back pain or discomfort from lying in the scanner. The noise from the scanner is loud enough to damage hearing, especially in people who already have hearing loss. Everyone having a research MRI scan will be fitted with hearing protection. If the hearing protection comes loose during the scan, you should let us know right away.

There are no known long-term risks of MRI scans.

o Risk for gadolinium enhanced MRI scans:

**Procedure:** During part of the MRI you may receive gadolinium, a contrast agent, through an intravenous (iv) catheter. It will be done for medical purposes.

It is not known if MRI with contrast is completely safe for a developing fetus. Therefore, all women of childbearing potential will have a pregnancy test performed no more than 24 hours before each MRI scan with contrast. The scan will not be done if the pregnancy test is positive.

**Risks:** The risks of an IV catheter include bleeding, infection, or inflammation of the skin and vein with pain and swelling.

Mild symptoms from gadolinium infusion occur in fewer than 1% of those who receive it and usually go away quickly. Mild symptoms may include coldness in the arm during the injection, a metallic taste, headache, and nausea. In an extremely small number, fewer than one in 300,000 people, more severe symptoms have been reported including shortness of breath, wheezing, hives, and lowering of blood pressure. You should not receive gadolinium if you previously had an allergic

## PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)




reaction to it. You will be asked about such allergic reactions before gadolinium is given.

People with kidney disease are at risk for a serious reaction to gadolinium contrast called "nephrogenic systemic fibrosis" which has resulted in a very small number of deaths. A blood test of your kidney function may be done within the month before an MRI scan with gadolinium contrast. You will not receive gadolinium for a research MRI scan if your kidney function is not normal or if you received gadolinium within the previous month.

Most of the gadolinium contrast leaves the body in the urine. However, the FDA recently issued a safety alert that indicates small amounts of gadolinium may remain in the body for months to years. The effects of the retained gadolinium are not clear. At this time, retained gadolinium has not been linked to health risks in people whose kidneys work well.

Some types of gadolinium contrast drugs are less likely to remain than others. In this study, we will use the gadolinium contrast drugs that are less likely to remain.

We will also give you additional information called a "Medication Guide." Upon request, we will give you individual information about retained gadolinium we see on your studies.

# What are the risks related to pregnancy?

You may not participate in this study if you are pregnant. If you are able to become pregnant, we will perform a pregnancy test before exposing you to radiation. You must tell us if you may have become pregnant within the previous 14 days because the pregnancy test is unreliable during that time.

#### What are the risks of radiation from being in the study?

During your participation in the screening portion of this study, you will be exposed to radiation from one CT scan of the chest, abdomen and pelvis and one 18F-FDG PET/CT. The amount of radiation exposure you will receive from these procedures is equal to approximately 2.3 rem. A rem is a unit of absorbed radiation.

Every day, people are exposed to low levels of radiation that come from the sun and the environment around them. The average person in the United States receives a radiation exposure of 0.3 rem per year from these sources. This type of radiation is called "background radiation." No one knows for sure whether exposure to these low amounts of radiation is harmful to your body.

The CT and PET scans that you get in this study will expose you to roughly the same amount of radiation as 7.7 years' worth of background radiation. Most of the time, this amount of extra radiation is not harmful to you. However, scientists believe that being exposed to too much radiation can cause harmful side effects. This could include getting a new cancer. We estimate that this could happen in about 1 out of every 1000 people who get a very large amount of extra radiation.

## PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)




## WHAT ARE THE BENEFITS OF BEING IN THE STUDY?

You might not benefit from being in this study.

This part of the study is only for screening. However, you may gain clinical information about your disease or your organ function that will be helpful to your overall medical care. This testing may make you eligible to participate in this research study at the NIH. You will also have the benefit of a consultation with one of the NIH doctors to discuss your treatment, and, if you so desire, the results of these screening tests and procedures will be communicated to your personal physician.

#### WHAT OTHER OPTIONS ARE THERE FOR YOU?

Before you decide whether or not to be in this study, we will discuss other options that are available to you. Instead of being in this study, you may choose not to be tested for eligibility or to have any other studies done.

## **DISCUSSION OF FINDINGS**

## New information about the study

If we find out any new information that may affect your choice to participate in this study, we will get in touch with you to explain what we have learned. This may be information we have learned while doing this study here at the NIH or information we have learned from other scientists doing similar research in other places.

## Return of research results

All of the clinical test results will be shared with you. We will discuss any findings that are abnormal with you. We can also share the findings of these screening evaluations with any medical provider that you wish to have this information.

#### EARLY WITHDRAWAL FROM THE STUDY

You will be removed from the study if:

• You are found not to be eligible for the study

You can stop taking part in the study at any time. However, if you decide to stop taking part in the study, we would like you to talk to the study doctor and your regular doctor first.

# STORAGE, SHARING AND FUTURE RESEARCH USING YOUR SPECIMENS AND DATA

## Will your specimens or data be saved for use in other research studies?

As part of this study, we are obtaining specimens and data from you. We will remove all the identifiers, such as your name, date of birth, address, or medical record number and label your specimens and data with a code so that you cannot easily be identified. However, the code will be linked through a key to information that can identify you. We plan to store and use these specimens and data for studies other than the ones described in this consent form that are going on right now, as well as studies that may be conducted in the future. These studies may provide additional information that will be helpful in understanding B-cell lymphoma, or other diseases or conditions. This could include studies to develop other research tests, treatments, drugs, or

## PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)




devices, that may lead to the development of a commercial product by the NIH and/or its research or commercial partners. There are no plans to provide financial compensation to you if this happens. Also, it is unlikely that we will learn anything from these studies that may directly benefit you.

I give permission for my coded specimens and data to be stored and used for future research as described above.

| Yes | No |
|----------|----------|
| Initials | Initials |

# Will your specimens or data be shared for use in other research studies?

We may share your coded specimens and data with other researchers. If we do, while we will maintain the code key, we will not share it, so the other researchers will not be able to identify you. They may be doing research in areas that are similar to this study or in other unrelated areas. These researchers may be at NIH, other research centers and institutions, or commercial entities.

I give permission for my coded specimens and data to be shared with other researchers and used by these researchers for future research as described above.

| Yes | No |
|----------|----------|
| Initials | Initials |

If you change your mind and do not want us to store and use your specimens and data for future research, you should contact the research team member identified at the top of this document. We will do our best to comply with your request but cannot guarantee that we will always be able to destroy your specimens and data. For example, if some research with your specimens and data has already been completed, the information from that research may still be used. Also, for example, if the specimens and data have been shared already with other researchers, it might not be possible to withdraw them.

In addition to the planned use and sharing described above, we might remove all identifiers and codes from your specimens and data and use or share them with other researchers for future research at the NIH or other places. When we or the other researchers access your anonymized data, there will be no way to link the specimens or data back to you. We will not contact you to ask your permission or otherwise inform you before we do this. We might do this even if you answered "no" to the above questions. If we do this, we would not be able to remove your specimens or data to prevent their use in future research studies, even if you asked, because we will not be able to tell which are your specimens or data.

## PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1) Version Date: 02/22/2023




NIH policies require that your clinical and other study data be placed in an internal NIH database that is accessible to other NIH researchers for future research. Usually, these researchers will not have access to any of your identifiers, such as your name, date of birth, address, or medical record number; and your data will be labeled with only a code. We cannot offer you a choice of whether your data to be placed in this database or not. If you do not wish to have your data placed in this database, you should not enroll in this study.

## How long will your specimens and data be stored by the NIH?

Your specimens and data may be stored by the NIH as long as the study is open. When this study is closed, we may keep the data and any samples that are leftover for future research indefinitely.

# Risks of storage and sharing of specimens and data

When we store your specimens and data, we take precautions to protect your information from others that should not have access to it. When we share your specimens and data, we will do everything we can to protect your identity, for example, when appropriate, we remove information that can identify you. Even with the safeguards we put in place, we cannot guarantee that your identity will never become known or someone may gain unauthorized access to your information. New methods may be created in the future that could make it possible to re-identify your specimens and data.

#### **PAYMENT**

# Will you receive any type of payment for taking part in this study?

You will not receive any payment for taking part in this study.

## REIMBURSEMENT

## Will you receive reimbursement or direct payment by NIH as part of your participation?

Some NIH Clinical Center studies offer reimbursement or payment for travel, lodging or meals while participating in the research. The amount, if any, is guided by NIH policies and guidelines.

On this study, the NCI will reimburse the cost for some of your expenses. Some of these costs may be paid directly by the NIH and some may be reimbursed after you have paid. The amount and form of these payments are determined by the NCI Travel and Lodging Reimbursement Policy. You will be given a summary of the policy which provides more information.

#### **COST**

# Will taking part in this research study cost you anything?

NIH does not bill health insurance companies or participants for any research or related clinical care that you receive at the NIH Clinical Center.

- If some tests and procedures are performed outside the NIH Clinical Center, you may have to pay for these costs if they are not covered by your insurance company.
- Medicines that are not part of the study treatment will not be provided or paid for by the NIH Clinical Center.
- Once you have completed taking part in the study, medical care will no longer be provided by the NIH Clinical Center.

## PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1) Version Date: 02/22/2023




## **CONFLICT OF INTEREST (COI)**

The National Institutes of Health (NIH) reviews NIH staff researchers at least yearly for conflicts of interest. This process is detailed in a COI Guide. You may ask your research team for a copy of the COI Guide or for more information. Members of the research team who do not work for NIH are expected to follow these guidelines or the guidelines of their home institution, but they do not need to report their personal finances to the NIH.

The NIH and the research team for this study are using a drug developed by Bayer Pharmaceuticals through a collaboration between your study team and the company. The company also provides financial support for this study.

## CLINICAL TRIAL REGISTRATION AND RESULTS REPORTING

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

## CONFIDENTIALITY PROTECTIONS PROVIDED IN THIS STUDY

Some of your health information, and/or information about your specimen, from this study will be kept in a central database for research. Your name or contact information will not be put in the database. Your test results will be identified by a unique code and the list that links the code to your name will be kept separate from your sample and health information. Your information may be given out if required by law. For example, certain states require doctors to report to health boards if they find a disease like tuberculosis. However, the researchers will do their best to make sure that any information that is released will not identify you.

# Will your medical information be kept private?

We will do our best to make sure that the personal information in your medical record will be kept private. However, we cannot guarantee total privacy. Organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

- The NIH and other government agencies, like the Food and Drug Administration (FDA), which are involved in keeping research safe for people.
- National Institutes of Health Intramural Institutional Review Board
- The study Sponsor, Center for Cancer Research or their agent(s)
- Qualified representatives from Bayer Pharmaceuticals, the pharmaceutical company who produces copanlisib.

The researchers conducting this study and the NIH follow applicable laws and policies to keep your identifying information private to the extent possible. However, there is always a chance that, despite our best efforts, your identity and/or information about your participation in this research may be inadvertently released or improperly accessed by unauthorized persons.

In most cases, the NIH will not release any identifiable information collected about you without your written permission. However, your information may be shared as described in the section of this document on sharing of specimens and data, and as further outlined in the following sections.

## PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)




Further, the information collected for this study is protected by NIH under a Certificate of Confidentiality and the Privacy Act.

# **Certificate of Confidentiality**

To help us protect your privacy, the NIH Intramural Program has received a Certificate of Confidentiality (Certificate). With this certificate, researchers may not release or use data or information about you except in certain circumstances.

NIH researchers must not share information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if requested by a court.

The Certificate does not protect your information when it:

- 1. is disclosed to people connected with the research, for example, information may be used for auditing or program evaluation internally by the NIH; or
- 2. is required to be disclosed by Federal, State, or local laws, for example, when information must be disclosed to meet the legal requirements of the federal Food and Drug Administration (FDA);
- 3. is for other research;
- 4. is disclosed with your consent.

The Certificate does not prevent you from voluntarily releasing information about yourself or your involvement in this research.

The Certificate will not be used to prevent disclosure to state or local authorities of harm to self or others including, for example, child abuse and neglect, and by signing below you consent to those disclosures. Other permissions for release may be made by signing NIH forms, such as the Notice and Acknowledgement of Information Practices consent.

## **Privacy Act**

The Federal Privacy Act generally protects the confidentiality of your NIH medical information that we collect under the authority of the Public Health Service Act. In some cases, the Privacy Act protections differ from the Certificate of Confidentiality. For example, sometimes the Privacy Act allows release of information from your record without your permission, for example, if it is requested by Congress. Information may also be released for certain research purposes with due consideration and protection, to those engaged by the agency for research purposes, to certain federal and state agencies, for HIV partner notification, for infectious disease or abuse or neglect reporting, to tumor registries, for quality assessment and medical audits, or when the NIH is involved in a lawsuit. However, NIH will only release information from your medical record if it is permitted by both the Certificate of Confidentiality and the Privacy Act.

## POLICY REGARDING RESEARCH-RELATED INJURIES

The NIH Clinical Center will provide short-term medical care for any injury resulting from your participation in research here. In general, no long-term medical care or financial compensation for research-related injuries will be provided by the NIH, the NIH Clinical Center, or the Federal Government. However, you have the right to pursue legal remedy if you believe that your injury justifies such action.

## PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)




## PROBLEMS OR QUESTIONS

If you have any problems or questions about this study, or about your rights as a research participant, or about any research-related injury, contact the Principal Investigator, Mark Roschewski, M.D., at mark.roschewski@nih.gov or 240-760-6183. You may also call the NIH Clinical Center Patient Representative at 301-496-2626, or the NIH Office of IRB Operations at 301-402-3713, if you have a research-related complaint or concern.

## **CONSENT DOCUMENT**

Please keep a copy of this document in case you want to read it again.

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1) Version Date: 02/22/2023




| Adult Research Participant: I have read the explanation about this study and have been given the opportunity to discuss it and to ask questions. I consent to participate in this study. | | |
|---|---|---|
| Signature of Research Participant | Print Name of Research Participant | Date |
| Investigator: | | |
| Signature of Investigator | Print Name of Investigator | Date |
| Witness should sign below if either: 1. A short form consent process has been used to enroll a non-English speaking subject or 2. An oral presentation of the full consent has been used to enroll a blind or illiterate subject Signature of Witness Print Name of Witness Date | | |
| 5 | | |
| NIH ADMINISTRATIVE SECTION TO BE COMPLETED REGARDING THE USE OF AN INTERPRETER: An interpreter, or other individual, who speaks English and the participant's preferred language facilitated | | |
| the administration of informed consent <u>and served as a witness</u> . The investigator obtaining consent may not also serve as the witness. | | |
| An interpreter, or other individual, who speaks English and the participant's preferred language facilitated the administration of informed consent but <u>did not</u> serve as a witness. The name or ID code of the person providing interpretive support is: | | |

PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


